CLINICAL TRIAL: NCT02072161
Title: A Randomized, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of ETC-1002 Versus Placebo in Patients With Hypercholesterolemia Receiving Ongoing Statin Therapy
Brief Title: Evaluation of ETC-1002 vs Placebo in Patients Receiving Ongoing Statin Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1002-009
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Hypercholesterolemia
Keywords: Statin; LDL; Cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ETC-1002 120 mg/day (Experimental): Orally, once daily in morning as capsules
  Interventions: Drug: ETC-1002; Drug: Statin Therapy
- ETC-1002 180 mg/day (Experimental): Orally, once daily in morning as capsules
  Interventions: Drug: ETC-1002; Drug: Statin Therapy
- Placebo (Placebo Comparator): Orally, once daily in morning
  Interventions: Drug: Placebo; Drug: Statin Therapy

INTERVENTIONS:
Drug: ETC-1002 — ETC-1002 capsules, taken once daily oral
  Arms: ETC-1002 120 mg/day; ETC-1002 180 mg/day
Drug: Placebo — Placebo capsules, taken once daily oral
  Arms: Placebo
Drug: Statin Therapy — Patients remained on ongoing statin therapy (not study provided) of either Atorvastatin 10mg or 20mg; Simvastatin 5mg, 10mg or 20mg; Rosuvastatin 5mg or 10mg; or Pravastatin 10mg, 20mg or 40mg.

SUMMARY:
The purpose of this research study is to see how ETC-1002 is tolerated in the body and how ETC-1002 affects the levels of LDL-C (bad cholesterol) in patients receiving ongoing statin therapy.

DETAILED DESCRIPTION:
Approximately 132 hypercholesterolemic patients already taking statin therapy to treat elevated LDL-C will be randomized in a ratio of 1:1:1 to receive either ETC-1002 (120 mg or 180 mg dose), or placebo for 12 weeks in addition to ongoing statin therapy. This study will explore the safety and efficacy of ETC-1002 when given to patients receiving statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Fasting, calculated mean LDL-C ≥130 mg/dL and ≤220 mg/dL
* Fasting mean TG level ≤400 mg/dL
* Stable statin therapy for at least 3 months prior to screening: atorvastatin (10 or 20 mg daily), simvastatin (5, 10 or 20 mg daily), rosuvastatin (5 or 10 mg daily), or pravastatin (10, 20 or 40 mg daily)

Exclusion Criteria:

* Clinically significant cardiovascular disease within 12 months of screening
* Current muscle-related symptoms that may be due to ongoing statin therapy or a history of certain lab abnormalities that occurred during statin therapy and resolved when statin therapy was discontinued
* Type 1 diabetes or uncontrolled type 2 diabetes
* Use of metformin or thiazolidinediones (TZD) within 4 weeks of screening
* History of chronic musculoskeletal symptoms such as fibromyalgia
* Uncontrolled hypothyroidism
* Liver disease or dysfunction
* Renal dysfunction or nephritic syndrome
* Gastrointestinal conditions or procedures or surgeries
* Hematologic or coagulation disorders or low hemoglobin levels
* HIV or AIDS
* History of malignancy
* History of drug or alcohol abuse within 2 years
* Use of experimental or investigational drugs within 30 days of screening
* Use of ETC-1002 in a previous clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in calculated low density lipoprotein-cholesterol (LDL-C) | 12 weeks

SECONDARY OUTCOMES:
Percent change in non-high-density lipoprotein cholesterol (non-HDL-C) | 12 weeks
Percent change in apolipoprotein B (ApoB) | 12 weeks
Percent change in total cholesterol (TC) | 12 weeks
Percent change in high-sensitivity C-reactive protein (hsCRP) | 12 weeks
Percent change in triglycerides (TG) | 12 weeks
Percent change in lipoprotein particle number | 12 weeks
Safety using adverse event reports; clinical laboratory results | 12 weeks
Safety using adverse event reports; vital signs | 12 weeks
Pharmacokinetic plasma trough concentrations of ETC-1002 and metabolite 15228 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diane E MacDougall, Study Director — Esperion Therapeutics, Inc.
Locations (39):
- United States (39):
  - Muscle Shoals, Alabama
  - Chandler, Arizona
  - Chino, California
  - Los Angeles, California
  - Sacramento, California
  - Walnut Creek, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Brandon, Florida
  - Jacksonville, Florida
  - Oviedo, Florida
  - Ponte Vedra, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Marietta, Georgia
  - Boise, Idaho
  - Meridian, Idaho
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Louisville, Kentucky
  - Port Gibson, Mississippi
  - Rochester, New York
  - Salisbury, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Franklin, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Tulsa, Oklahoma
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Summerville, South Carolina
  - Kingsport, Tennessee
  - Houston, Texas
  - Bountiful, Utah
  - Orem, Utah
  - Norfolk, Virginia
  - Richmond, Virginia

REFERENCES:
- [Background] Gutierrez MJ, Rosenberg NL, Macdougall DE, Hanselman JC, Margulies JR, Strange P, Milad MA, McBride SJ, Newton RS. Efficacy and safety of ETC-1002, a novel investigational low-density lipoprotein-cholesterol-lowering therapy for the treatment of patients with hypercholesterolemia and type 2 diabetes mellitus. Arterioscler Thromb Vasc Biol. 2014 Mar;34(3):676-83. doi: 10.1161/ATVBAHA.113.302677. Epub 2014 Jan 2. PMID 24385236
- [Background] Ballantyne CM, Davidson MH, Macdougall DE, Bays HE, Dicarlo LA, Rosenberg NL, Margulies J, Newton RS. Efficacy and safety of a novel dual modulator of adenosine triphosphate-citrate lyase and adenosine monophosphate-activated protein kinase in patients with hypercholesterolemia: results of a multicenter, randomized, double-blind, placebo-controlled, parallel-group trial. J Am Coll Cardiol. 2013 Sep 24;62(13):1154-62. doi: 10.1016/j.jacc.2013.05.050. Epub 2013 Jun 13. PMID 23770179
- [Background] Filippov S, Pinkosky SL, Lister RJ, Pawloski C, Hanselman JC, Cramer CT, Srivastava RAK, Hurley TR, Bradshaw CD, Spahr MA, Newton RS. ETC-1002 regulates immune response, leukocyte homing, and adipose tissue inflammation via LKB1-dependent activation of macrophage AMPK. J Lipid Res. 2013 Aug;54(8):2095-2108. doi: 10.1194/jlr.M035212. Epub 2013 May 24. PMID 23709692
- [Background] Pinkosky SL, Filippov S, Srivastava RA, Hanselman JC, Bradshaw CD, Hurley TR, Cramer CT, Spahr MA, Brant AF, Houghton JL, Baker C, Naples M, Adeli K, Newton RS. AMP-activated protein kinase and ATP-citrate lyase are two distinct molecular targets for ETC-1002, a novel small molecule regulator of lipid and carbohydrate metabolism. J Lipid Res. 2013 Jan;54(1):134-51. doi: 10.1194/jlr.M030528. Epub 2012 Nov 1. PMID 23118444